CLINICAL TRIAL: NCT03166813
Title: Remote Ischaemic Preconditioning in Paediatric Cancer Patients Receiving Anthracycline Therapy
Brief Title: Remote Ischaemic Preconditioning in Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yiu-fai Cheung, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW17-143
Record Dates: First submitted 2017-05-16; First posted 2017-05-25 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Cardiotoxicity
Keywords: remote ischaemic preconditioning; childhood cancer; cardio-oncology; anthracycline; myocardial reperfusion injury
MeSH Terms: conditions — Cardiotoxicity; Neoplasms; Myocardial Reperfusion Injury | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention RIPC (Experimental): The intervention RIPC protocol will be induced by three cycles of inflation of a blood pressure cuff placed over the upper or lower limb, where deemed to cause minimal discomfort to patient, to 15 mmHg above the systolic blood pressure for five minutes followed by five minutes of cuff deflation to 0 mmHg.
  Interventions: Procedure: Remote Ischaemic Preconditioning
- Control (Placebo Comparator): The control protocol involves only placement of blood pressure cuff but without inflation for 30 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Remote Ischaemic Preconditioning — The intervention RIPC protocol will be performed each time by three cycles of inflation of a blood pressure cuff placed over the arm or leg of your child, where deemed to cause minimal discomfort, to 15 mmHg above the systolic blood pressure for 5 minutes followed by 5 minutes of cuff deflation to 0 mmHg.
  Other Names: Remote Ischemic Conditioning; Remote Ischaemic Conditioning
  Arms: Intervention RIPC
Other: Control — Placement of blood pressure cuff without inflation for 30 minutes.
  Other Names: Sham
  Arms: Control

SUMMARY:
Survival rates of children with cancers have improved significantly in the recent few decades. Nonetheless, the side effect of this class of drugs on heart function remains to be an issue of concern. Exploration of new strategies to protect the heart in the long term is therefore of paramount importance in children undergoing treatment of cancers. Previous cardioprotective interventions hav focused on changing the formulation or rate of administration of anthracyclines but with no observable benefits. While dexrazoxane, an iron chelator, has shown to reduce cardiotoxic outcomes, there remains worries of an association between dexrazoxane use and an increased risk of developing secondary malignancies. Recently, the clinical application of remote ischaemic preconditioning (RIPC) as a non-invasive and an easily applicable non-pharmacological myocardial protective intervention has gained increasing interest. Remote ischaemic preconditioning is the phenomenon in which brief episodes of reversible ischaemia and reperfusion applied to one vascular bed render resistance to ischaemia reperfusion injury of tissues and organs distant away. It can be achieved by repeated 5-minute cycles of inflation and deflation of blood pressure cuff placed over the arm or leg to induce limb ischaemia and reperfusion injury. It is noteworthy that anthracycline cardiotoxicity and myocardial reperfusion injury occur through similar pathways. Hence, the investigators hypothesize that RIPC may reduce myocardial injury in children receiving anthracycline chemotherapy for childhood malignancies. The proposed study aims to conduct a parallel-group blinded randomized controlled trial study to investigate whether RIPC may reduce heart damage in childhood cancer patients undergoing anthracycline-based treatment, and to determine the effect of RIPC on the changes in levels of cardiac troponin T, and on the occurrence of clinical cardiovascular events and echocardiographic indices.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) protocol will be induced at baseline and before each dose of anthracycline cardiac surgery and once before induction of anesthesia by 3 cycles of 5-min upper or lower limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to 15 mmHg above the systolic blood pressure for 5 minutes followed by 5 minutes of cuff deflation to 0 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 4 to 18 years old
* newly diagnosed patients with solid tumours or haematological malignancies referred for anthracycline-based chemotherapy
* no history of being treated with anthracycline-based regimens in the past.

Exclusion Criteria:

* existence of congenital or acquired heart disease
* presence of syndromal disorders
* abnormal baseline echocardiographic assessment
* peripheral vascular disease that renders RIPC impossible
* a platelet count <30,000/µL.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
High sensitivity cardiac troponin T (hs-cTnT) | hs-cTnT will be measured at baseline, and at 3 months after completion of all anthracycline. The change from baseline hs-cTnT to at 3 months after completion of all anthracycline will be measured.
  Biomarker of myocardial injury

SECONDARY OUTCOMES:
Occurrence of clinical cardiovascular events | at baseline, within 1 week and at 3 months after completion of all anthracycline treatment.
  Clinical cardiovascular events include development of clinical congestive heart failure, occurrence of cardiac arrhythmias, the need to institute cardiac medications, and cardiac death
Echocardiographic assessment of left ventricular function | Echocardiographic assessment will be performed at baseline, and within 1 week and at 3 months after completion of all anthracycline treatment.
  left ventricular systolic and diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Yiu-fai Cheung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Candilio L, Malik A, Ariti C, Barnard M, Di Salvo C, Lawrence D, Hayward M, Yap J, Roberts N, Sheikh A, Kolvekar S, Hausenloy DJ, Yellon DM. Effect of remote ischaemic preconditioning on clinical outcomes in patients undergoing cardiac bypass surgery: a randomised controlled clinical trial. Heart. 2015 Feb;101(3):185-92. doi: 10.1136/heartjnl-2014-306178. Epub 2014 Sep 24. PMID 25252696
- [Background] Venugopal V, Hausenloy DJ, Ludman A, Di Salvo C, Kolvekar S, Yap J, Lawrence D, Bognolo J, Yellon DM. Remote ischaemic preconditioning reduces myocardial injury in patients undergoing cardiac surgery with cold-blood cardioplegia: a randomised controlled trial. Heart. 2009 Oct;95(19):1567-71. doi: 10.1136/hrt.2008.155770. Epub 2009 Jun 8. PMID 19508973
- [Background] Chung R, Maulik A, Hamarneh A, Hochhauser D, Hausenloy DJ, Walker JM, Yellon DM. Effect of Remote Ischaemic Conditioning in Oncology Patients Undergoing Chemotherapy: Rationale and Design of the ERIC-ONC Study--A Single-Center, Blinded, Randomized Controlled Trial. Clin Cardiol. 2016 Feb;39(2):72-82. doi: 10.1002/clc.22507. Epub 2016 Jan 25. PMID 26807534
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Background] McCrindle BW, Clarizia NA, Khaikin S, Holtby HM, Manlhiot C, Schwartz SM, Caldarone CA, Coles JG, Van Arsdell GS, Scherer SW, Redington AN. Remote ischemic preconditioning in children undergoing cardiac surgery with cardiopulmonary bypass: a single-center double-blinded randomized trial. J Am Heart Assoc. 2014 Jul 28;3(4):e000964. doi: 10.1161/JAHA.114.000964. PMID 25074698
- [Derived] Cheung YF, Li VW, So EK, Cheng FW, Yau JP, Chiu SY, Wong WH, Cheuk DK. Remote Ischemic Conditioning in Pediatric Cancer Patients Receiving Anthracycline Chemotherapy: A Sham-Controlled Single-Blind Randomized Trial. JACC CardioOncol. 2023 Mar 21;5(3):332-342. doi: 10.1016/j.jaccao.2022.11.020. eCollection 2023 Jun. PMID 37397078